CLINICAL TRIAL: NCT06446622
Title: Influence of Biological Sex and Age on Cerebral Blood Flow and Vessel Function During Exercise: a Pilot Study
Brief Title: Brain Blood Flow Responses During Exercise: Younger Cohort
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-0512: Younger Cohort; Protocol Version 3/22/2023 (Other: UW Madison); A176000 (Other: UW Madison); UWF (Other: University of Wisconsin Foundation)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cerebrovascular Circulation; Magnetic Resonance Imaging
Keywords: Magnetic Resonance Imaging; Exercise; Brain Blood Flow
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Young Adults (Experimental): Young Adults between 20-40 years of age.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Participants will undergo an MRI scan while performing exercise at two intensities (light and moderate/vigorous) using an MRI-compatible stepper device.

SUMMARY:
Brain blood flow will be measured during exercise using magnetic resonance imaging.

DETAILED DESCRIPTION:
Over 6 million Americans are living with Alzheimer's disease and related dementias and this number is expected to reach over 13 million by 2060. Thus, there is an urgent need for interventions to prevent the development and progression of Alzheimer's disease and related dementias. Regular exercise is currently the most promising strategy as it is repeatedly shown to have neuroprotective benefits. Evidence suggests that the neuroprotective effects of exercise is the result of improved health of blood vessels. Despite the vast amount of evidence on the benefit of exercise on the peripheral vasculature, there is little information regarding brain vascular responses during exercise. This study will investigate the impact of exercise at varying intensities on brain blood flow during exercise, and will also examine the influence of age and sex.

This record represents a younger cohort for the study represented in NCT05864950.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 20-40 years old
* Demonstrate an exercise history of engaging in aerobic physical activity at least 3 times per week for a minimum of 30 continuous minutes
* Have experience using cardiovascular exercise equipment (e.g., treadmill, elliptical, upright or recumbent bicycle, stair-stepper)

Exclusion Criteria:

* Outside of specified age range
* Do not have experience using cardiovascular exercise equipment
* Do not meet the physical activity criteria
* Present with a history or evidence of hepatic, renal, hematological disease, cardiovascular disease including uncontrolled hypertension, peripheral vascular disease, stroke/neurovascular disease, and diabetes
* have a body mass index ≥35 kg/m2
* are ≥ 71 inches (180 cm) in height
* have any contraindications to MRI
* currently use or have a history of use of tobacco or illegal substances
* have current and/or a history of depression or other mood related disorders (those with mild depression and/or anxiety that is controlled with medication and/or therapy will not be excluded)
* vulnerable populations (e.g., pregnant women, prisoners, individuals lacking capacity to consent)
* if the desired moderate/vigorous exercise intensity corresponds to > 350 watts on the stepper device

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cerebral Hemodynamics | One study visit, up to 120 minutes
  The change in cross-sectional area of the cerebral arteries during exercise will be measured with MRI.
Cerebral Blood Flow | One study visit, up to 120 minutes
  The change in intracranial blood flow during exercise will be measured with MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matthews KA, Xu W, Gaglioti AH, Holt JB, Croft JB, Mack D, McGuire LC. Racial and ethnic estimates of Alzheimer's disease and related dementias in the United States (2015-2060) in adults aged >/=65 years. Alzheimers Dement. 2019 Jan;15(1):17-24. doi: 10.1016/j.jalz.2018.06.3063. Epub 2018 Sep 19. PMID 30243772
- [Background] Barnes JN, Corkery AT. Exercise Improves Vascular Function, but does this Translate to the Brain? Brain Plast. 2018 Dec 12;4(1):65-79. doi: 10.3233/BPL-180075. PMID 30564547
- [Background] Mitchell GF. Effects of central arterial aging on the structure and function of the peripheral vasculature: implications for end-organ damage. J Appl Physiol (1985). 2008 Nov;105(5):1652-60. doi: 10.1152/japplphysiol.90549.2008. Epub 2008 Sep 4. PMID 18772322
- [Background] Silvestrini M, Pasqualetti P, Baruffaldi R, Bartolini M, Handouk Y, Matteis M, Moffa F, Provinciali L, Vernieri F. Cerebrovascular reactivity and cognitive decline in patients with Alzheimer disease. Stroke. 2006 Apr;37(4):1010-5. doi: 10.1161/01.STR.0000206439.62025.97. Epub 2006 Feb 23. PMID 16497984
- [Background] Vicenzini E, Ricciardi MC, Altieri M, Puccinelli F, Bonaffini N, Di Piero V, Lenzi GL. Cerebrovascular reactivity in degenerative and vascular dementia: a transcranial Doppler study. Eur Neurol. 2007;58(2):84-9. doi: 10.1159/000103642. Epub 2007 Jun 12. PMID 17565221
- [Background] Rubanyi GM, Romero JC, Vanhoutte PM. Flow-induced release of endothelium-derived relaxing factor. Am J Physiol. 1986 Jun;250(6 Pt 2):H1145-9. doi: 10.1152/ajpheart.1986.250.6.H1145. PMID 3487253
- [Background] Harvey PJ, Picton PE, Su WS, Morris BL, Notarius CF, Floras JS. Exercise as an alternative to oral estrogen for amelioration of endothelial dysfunction in postmenopausal women. Am Heart J. 2005 Feb;149(2):291-7. doi: 10.1016/j.ahj.2004.08.036. PMID 15846267
- [Background] Black MA, Cable NT, Thijssen DH, Green DJ. Impact of age, sex, and exercise on brachial artery flow-mediated dilatation. Am J Physiol Heart Circ Physiol. 2009 Sep;297(3):H1109-16. doi: 10.1152/ajpheart.00226.2009. Epub 2009 Jul 24. PMID 19633208
- [Background] Duckles SP, Miller VM. Hormonal modulation of endothelial NO production. Pflugers Arch. 2010 May;459(6):841-51. doi: 10.1007/s00424-010-0797-1. Epub 2010 Mar 7. PMID 20213497
- [Background] Moreau KL, Stauffer BL, Kohrt WM, Seals DR. Essential role of estrogen for improvements in vascular endothelial function with endurance exercise in postmenopausal women. J Clin Endocrinol Metab. 2013 Nov;98(11):4507-15. doi: 10.1210/jc.2013-2183. Epub 2013 Oct 3. PMID 24092827
- [Background] Miller KB, Howery AJ, Rivera-Rivera LA, Johnson SC, Rowley HA, Wieben O, Barnes JN. Age-Related Reductions in Cerebrovascular Reactivity Using 4D Flow MRI. Front Aging Neurosci. 2019 Oct 17;11:281. doi: 10.3389/fnagi.2019.00281. eCollection 2019. PMID 31680935
- [Background] Ogoh S, Ainslie PN. Cerebral blood flow during exercise: mechanisms of regulation. J Appl Physiol (1985). 2009 Nov;107(5):1370-80. doi: 10.1152/japplphysiol.00573.2009. Epub 2009 Sep 3. PMID 19729591
- [Background] Soucy KG, Ryoo S, Benjo A, Lim HK, Gupta G, Sohi JS, Elser J, Aon MA, Nyhan D, Shoukas AA, Berkowitz DE. Impaired shear stress-induced nitric oxide production through decreased NOS phosphorylation contributes to age-related vascular stiffness. J Appl Physiol (1985). 2006 Dec;101(6):1751-9. doi: 10.1152/japplphysiol.00138.2006. PMID 17106067
- [Background] Smith KJ, Ainslie PN. Regulation of cerebral blood flow and metabolism during exercise. Exp Physiol. 2017 Nov 1;102(11):1356-1371. doi: 10.1113/EP086249. Epub 2017 Sep 30. PMID 28786150
- [Background] Smith KJ, Wong LE, Eves ND, Koelwyn GJ, Smirl JD, Willie CK, Ainslie PN. Regional cerebral blood flow distribution during exercise: influence of oxygen. Respir Physiol Neurobiol. 2012 Oct 15;184(1):97-105. doi: 10.1016/j.resp.2012.07.014. Epub 2012 Aug 16. PMID 22926137
- [Background] Ogoh S, Tsukamoto H, Hirasawa A, Hasegawa H, Hirose N, Hashimoto T. The effect of changes in cerebral blood flow on cognitive function during exercise. Physiol Rep. 2014 Sep 28;2(9):e12163. doi: 10.14814/phy2.12163. Print 2014 Sep 1. PMID 25263210
- [Background] Caldwell HG, Coombs GB, Howe CA, Hoiland RL, Patrician A, Lucas SJE, Ainslie PN. Evidence for temperature-mediated regional increases in cerebral blood flow during exercise. J Physiol. 2020 Apr;598(8):1459-1473. doi: 10.1113/JP278827. Epub 2020 Feb 6. PMID 31912506
- [Background] Macdonald JA, Beshish AG, Corrado PA, Barton GP, Goss KN, Eldridge MW, Francois CJ, Wieben O. Feasibility of Cardiovascular Four-dimensional Flow MRI during Exercise in Healthy Participants. Radiol Cardiothorac Imaging. 2020 Jun 18;2(3):e190033. doi: 10.1148/ryct.2020190033. PMID 32734274
- [Background] Macdonald JA, Roberts GS, Corrado PA, Beshish AG, Haraldsdottir K, Barton GP, Goss KN, Eldridge MW, Francois CJ, Wieben O. Exercise-induced irregular right heart flow dynamics in adolescents and young adults born preterm. J Cardiovasc Magn Reson. 2021 Oct 21;23(1):116. doi: 10.1186/s12968-021-00816-2. PMID 34670573
- [Background] Miller KB, Gallo SJ, Rivera-Rivera LA, Corkery AT, Howery AJ, Johnson SC, Rowley HA, Wieben O, Barnes JN. Vertebral artery hypoplasia influences age-related differences in blood flow of the large intracranial arteries. Aging Brain. 2021 Jun 24;1:100019. doi: 10.1016/j.nbas.2021.100019. eCollection 2021. PMID 36911510
- [Background] Barnes JN. Exercise, cognitive function, and aging. Adv Physiol Educ. 2015 Jun;39(2):55-62. doi: 10.1152/advan.00101.2014. PMID 26031719
- [Background] Ferretti MT, Iulita MF, Cavedo E, Chiesa PA, Schumacher Dimech A, Santuccione Chadha A, Baracchi F, Girouard H, Misoch S, Giacobini E, Depypere H, Hampel H; Women's Brain Project and the Alzheimer Precision Medicine Initiative. Sex differences in Alzheimer disease - the gateway to precision medicine. Nat Rev Neurol. 2018 Aug;14(8):457-469. doi: 10.1038/s41582-018-0032-9. PMID 29985474
- [Background] Beam CR, Kaneshiro C, Jang JY, Reynolds CA, Pedersen NL, Gatz M. Differences Between Women and Men in Incidence Rates of Dementia and Alzheimer's Disease. J Alzheimers Dis. 2018;64(4):1077-1083. doi: 10.3233/JAD-180141. PMID 30010124
- See also: Brain Blood Flow Responses During Exercise - Older Cohort — https://clinicaltrials.gov/study/NCT05864950